CLINICAL TRIAL: NCT04215939
Title: Assessment of Vasomotion of People With Spinal Cord Injury
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Petros Dinas (Other)
Collaborators: European Commission (Other)
Responsible Party: Sponsor-Investigator, Petros Dinas, Senior Researcher in human physiology, University of Thessaly
Organization: University of Thessaly (Other)
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: 9. Vasomotion & spinal
Record Dates: First submitted 2019-12-30; First posted 2020-01-02 (Actual); Last update posted 2020-11-04 (Actual); Status verified 2020-11

CONDITIONS: Spinal Cord Injuries; Paraplegia
Keywords: Spinal cord injury; vasomotion; core temperature; sudomotor; thermoregulation
MeSH Terms: conditions — Spinal Cord Injuries; Paraplegia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (9):
- Cold environment participants with spinal cord injury (Experimental): In a cold environment (15-17°C and 40-50% relative humidity), participants will stay in a sited position for 20 minutes in order to collect baseline data and to allow their blood flow and body temperature adapt to the exposing environmental condition. Immediately after the baseline period participants will immerse their left hand and foot in warm water (34-36°C) for five minutes for a consistent starting (hand and foot) temperature. Following that participants will immerse their hand and foot in cold water (8°C) for 40 minutes.
  Interventions: Behavioral: Cold environment participants with spinal cord injury; Behavioral: Cold environment healthy male participants; Behavioral: Cold environment healthy female participants
- Thermoneutral environment participants with spinal cord injury (Experimental): In a thermoneutral enviroment (22-24°C and 40-50% relative humidity), participants will stay in a sited position for 20 minutes in order to collect baseline data and to allow their blood flow and body temperature adapt to the exposing environmental condition. Immediately after the baseline period participants will immerse their left hand and foot in warm water (34-36°C) for five minutes for a consistent starting (hand and foot) temperature. Following that participants will immerse their hand and foot in cold water (8°C) for 40 minutes.
  Interventions: Behavioral: Thermoneutral environment participants with spinal cord injury; Behavioral: Thermoneutral environment healthy male participants; Behavioral: Thermoneutral environment healthy female participants
- Warm environment participants with spinal cord injury (Experimental): In a warm environment (33-35°C and 40-50% relative humidity), participants will stay in a sited position for 20 minutes in order to collect baseline data and to allow their blood flow and body temperature adapt to the exposing environmental condition. Immediately after the baseline period participants will immerse their left hand and foot in warm water (34-36°C) for five minutes for a consistent starting (hand and foot) temperature. Following that participants will immerse their hand and foot in cold water (8°C) for 40 minutes.
  Interventions: Behavioral: Warm environment participants with spinal cord injury; Behavioral: Warm environment healthy male participants; Behavioral: Warm environment healthy female participants
- Cold environment healthy male participants (Active Comparator): In a cold environment (15-17°C and 40-50% relative humidity), participants will stay in a sited position for 20 minutes in order to collect baseline data and to allow their blood flow and body temperature adapt to the exposing environmental condition. Immediately after the baseline period participants will immerse their left hand and foot in warm water (34-36°C) for five minutes for a consistent starting (hand and foot) temperature. Following that participants will immerse their hand and foot in cold water (8°C) for 40 minutes.
  Interventions: Behavioral: Cold environment participants with spinal cord injury; Behavioral: Cold environment healthy male participants; Behavioral: Cold environment healthy female participants
- Thermoneutral environment healthy male participants (Active Comparator): In a thermoneutral enviroment (22-24°C and 40-50% relative humidity), participants will stay in a sited position for 20 minutes in order to collect baseline data and to allow their blood flow and body temperature adapt to the exposing environmental condition. Immediately after the baseline period participants will immerse their left hand and foot in warm water (34-36°C) for five minutes for a consistent starting (hand and foot) temperature. Following that participants will immerse their hand and foot in cold water (8°C) for 40 minutes.
  Interventions: Behavioral: Thermoneutral environment participants with spinal cord injury; Behavioral: Thermoneutral environment healthy male participants; Behavioral: Thermoneutral environment healthy female participants
- Warm environment healthy male participants (Active Comparator): In a warm environment (33-35°C and 40-50% relative humidity), participants will stay in a sited position for 20 minutes in order to collect baseline data and to allow their blood flow and body temperature adapt to the exposing environmental condition. Immediately after the baseline period participants will immerse their left hand and foot in warm water (34-36°C) for five minutes for a consistent starting (hand and foot) temperature. Following that participants will immerse their hand and foot in cold water (8°C) for 40 minutes.
  Interventions: Behavioral: Warm environment participants with spinal cord injury; Behavioral: Warm environment healthy male participants; Behavioral: Warm environment healthy female participants
- Cold environment healthy female participants (Active Comparator): In a cold environment (15-17°C and 40-50% relative humidity), participants will stay in a sited position for 20 minutes in order to collect baseline data and to allow their blood flow and body temperature adapt to the exposing environmental condition. Immediately after the baseline period participants will immerse their left hand and foot in warm water (34-36°C) for five minutes for a consistent starting (hand and foot) temperature. Following that participants will immerse their hand and foot in cold water (8°C) for 40 minutes.
  Interventions: Behavioral: Cold environment participants with spinal cord injury; Behavioral: Cold environment healthy male participants; Behavioral: Cold environment healthy female participants
- Thermoneutral environment healthy female participants (Active Comparator): In a thermoneutral enviroment (22-24°C and 40-50% relative humidity), participants will stay in a sited position for 20 minutes in order to collect baseline data and to allow their blood flow and body temperature adapt to the exposing environmental condition. Immediately after the baseline period participants will immerse their left hand and foot in warm water (34-36°C) for five minutes for a consistent starting (hand and foot) temperature. Following that participants will immerse their hand and foot in cold water (8°C) for 40 minutes.
  Interventions: Behavioral: Thermoneutral environment participants with spinal cord injury; Behavioral: Thermoneutral environment healthy male participants
- Warm enviroment healthy fmale participants (Active Comparator): In a warm environment (33-35°C and 40-50% relative humidity), participants will stay in a sited position for 20 minutes in order to collect baseline data and to allow their blood flow and body temperature adapt to the exposing environmental condition. Immediately after the baseline period participants will immerse their left hand and foot in warm water (34-36°C) for five minutes for a consistent starting (hand and foot) temperature. Following that participants will immerse their hand and foot in cold water (8°C) for 40 minutes.
  Interventions: Behavioral: Warm environment participants with spinal cord injury; Behavioral: Warm environment healthy male participants; Behavioral: Warm environment healthy female participants

INTERVENTIONS:
Behavioral: Cold environment participants with spinal cord injury — In a cold environment (15-17°C and 40-50% relative humidity), participants will stay in a sited position for 20 minutes in order to collect baseline data and to allow their blood flow and body temperature adapt to the exposing environmental condition. Immediately after the baseline period participants will immerse their left hand and foot in warm water (34-36°C) for five minutes for a consistent starting (hand and foot) temperature. Following that participants will immerse their hand and foot in cold water (8°C) for 40 minutes.
  Arms: Cold environment healthy female participants; Cold environment healthy male participants; Cold environment participants with spinal cord injury
Behavioral: Thermoneutral environment participants with spinal cord injury — In a thermoneutral environment (22-24°C and 40-50% relative humidity), participants will stay in a sited position for 20 minutes in order to collect baseline data and to allow their blood flow and body temperature adapt to the exposing environmental condition. Immediately after the baseline period participants will immerse their left hand and foot in warm water (34-36°C) for five minutes for a consistent starting (hand and foot) temperature. Following that participants will immerse their hand and foot in cold water (8°C) for 40 minutes.
  Arms: Thermoneutral environment healthy female participants; Thermoneutral environment healthy male participants; Thermoneutral environment participants with spinal cord injury
Behavioral: Warm environment participants with spinal cord injury — In a warm environment (33-35°C and 40-50% relative humidity), participants will stay in a sited position for 20 minutes in order to collect baseline data and to allow their blood flow and body temperature adapt to the exposing environmental condition. Immediately after the baseline period participants will immerse their left hand and foot in warm water (34-36°C) for five minutes for a consistent starting (hand and foot) temperature. Following that participants will immerse their hand and foot in cold water (8°C) for 40 minutes.
  Arms: Warm enviroment healthy fmale participants; Warm environment healthy male participants; Warm environment participants with spinal cord injury
Behavioral: Cold environment healthy male participants — In a cold environment (15-17°C and 40-50% relative humidity), participants will stay in a sited position for 20 minutes in order to collect baseline data and to allow their blood flow and body temperature adapt to the exposing environmental condition. Immediately after the baseline period participants will immerse their left hand and foot in warm water (34-36°C) for five minutes for a consistent starting (hand and foot) temperature. Following that participants will immerse their hand and foot in cold water (8°C) for 40 minutes.
  Arms: Cold environment healthy female participants; Cold environment healthy male participants; Cold environment participants with spinal cord injury
Behavioral: Thermoneutral environment healthy male participants — In a thermoneutral environment (22-24°C and 40-50% relative humidity), participants will stay in a sited position for 20 minutes in order to collect baseline data and to allow their blood flow and body temperature adapt to the exposing environmental condition. Immediately after the baseline period participants will immerse their left hand and foot in warm water (34-36°C) for five minutes for a consistent starting (hand and foot) temperature. Following that participants will immerse their hand and foot in cold water (8°C) for 40 minutes.
  Arms: Thermoneutral environment healthy female participants; Thermoneutral environment healthy male participants; Thermoneutral environment participants with spinal cord injury
Behavioral: Warm environment healthy male participants — In a warm environment (33-35°C and 40-50% relative humidity), participants will stay in a sited position for 20 minutes in order to collect baseline data and to allow their blood flow and body temperature adapt to the exposing environmental condition. Immediately after the baseline period participants will immerse their left hand and foot in warm water (34-36°C) for five minutes for a consistent starting (hand and foot) temperature. Following that participants will immerse their hand and foot in cold water (8°C) for 40 minutes.
  Arms: Warm enviroment healthy fmale participants; Warm environment healthy male participants; Warm environment participants with spinal cord injury
Behavioral: Cold environment healthy female participants — In a cold environment (15-17°C and 40-50% relative humidity), participants will stay in a sited position for 20 minutes in order to collect baseline data and to allow their blood flow and body temperature adapt to the exposing environmental condition. Immediately after the baseline period participants will immerse their left hand and foot in warm water (34-36°C) for five minutes for a consistent starting (hand and foot) temperature. Following that participants will immerse their hand and foot in cold water (8°C) for 40 minutes.
  Arms: Cold environment healthy female participants; Cold environment healthy male participants; Cold environment participants with spinal cord injury
Behavioral: Thermoneutral environment healthy female participants — In a thermoneutral environment (22-24°C and 40-50% relative humidity), participants will stay in a sited position for 20 minutes in order to collect baseline data and to allow their blood flow and body temperature adapt to the exposing environmental condition. Immediately after the baseline period participants will immerse their left hand and foot in warm water (34-36°C) for five minutes for a consistent starting (hand and foot) temperature. Following that participants will immerse their hand and foot in cold water (8°C) for 40 minutes.
  Arms: Thermoneutral environment healthy male participants; Thermoneutral environment participants with spinal cord injury
Behavioral: Warm environment healthy female participants — In a warm environment (33-35°C and 40-50% relative humidity), participants will stay in a sited position for 20 minutes in order to collect baseline data and to allow their blood flow and body temperature adapt to the exposing environmental condition. Immediately after the baseline period participants will immerse their left hand and foot in warm water (34-36°C) for five minutes for a consistent starting (hand and foot) temperature. Following that participants will immerse their hand and foot in cold water (8°C) for 40 minutes.
  Arms: Warm enviroment healthy fmale participants; Warm environment healthy male participants; Warm environment participants with spinal cord injury

SUMMARY:
Spinal cord injury (SCI), causes loss of supra-spinal control of the sympathetic nervous system and in some cases loss of sensation. As a result, people with SCI have impaired thermoregulatory system and the consequence of this thermoregulatory dysfunction, is that they cannot respond to the environmental changes. All the above lead to dysregulation in vasomotor tone, skeletal muscle shivering and sweating dysfunction. It is well known that skin plays an important role in regulating body temperature and regulates interactions between the environment and human body. A previous study in people with incomplete SCI showed that there are no differences in core temperature between patients with different level of mobility and sensation and different level of lesion, but there are significant differences in skin temperature. As mentioned above people with SCI have an impaired thermoregulatory capacity due to sudomotor and vasomotor dysfunction and that leads to greater thermal strain during rest and exercise when they expose to hot conditions. A previous study that performed exercise in people with SCI, highlights the fact that because of the impaired evaporative heat loss during exercise in hot conditions, they are in great risk. Because of this risk they propose different cooling strategies that promote evaporation such as fans and water spraying. It is therefore important to observe the thermoregulatory function (vasomotion and sudomotor) in people with SCI when they are exposed to different environments (cold, neutral and warm).

DETAILED DESCRIPTION:
The participants will visit the laboratory three times. At each time the environmental chamber will simulate a different environment in a random order for each participant. The three different environments will be as follow:

1. Cold environment 15-17°C and 40-50% relative humidity
2. Thermoneutral environment 22-24°C and 40-50% relative humidity
3. Warm environment 33-35°C and 40-50% relative humidity The participants will stay in a sited position for 20 minutes in order to collect baseline data and to allow to their blood flow and body temperature adapt to the exposing environmental condition each time. Immediately after the baseline period the participants will immerse their left hand and foot in warm water (34-36°C) for 5 minutes for a consistent starting (hand and foot) temperature. Following that participants will immerse their hand and foot in cold water (8°C) for 40 minutes. This procedure will be repeated in every measurement and it will only change the environment.

Anthropometric data [self-reported age, self-reported body stature and body mass (DXA, Lunar, GE Healthcare Boston, Massachusetts, U.S)] will be collecting at the beginning of the first measurement. Medical history of all the participants will be recording. During the study, continuous heart rate (Polar Team2. Polar Electro Oy, Kempele, Finland), core temperature (telemetric capsules BodyCap, Caen, France), mean skin temperature (wireless thermistors iButtons type DS1921H, Maxim/Dallas Semiconductor Corp., USA), finger temperature ((Smartreader 8 Plus, ACR, Vancouver, Canada), skin blood flow and sweat rate data (laser Doppler flow-meter PeriFlux System 5010, function unit; Perimed, Stockholm, Sweden and PeriFlux System 4002, master unit, satellite unit; Perimed, Stockholm, Sweden) will be collecting. Blood pressure will also be monitoring every 10 minutes with an automatic sphygmomanometer (Omron Healthcare M6 comfort, Japan). Skin temperature data will be collecting from four sites (chest, arm, thigh, and leg) and will be expressed as mean skin temperature according to the formula of Ramanathan (Tsk = [0.3(chest + arm) + 0.2(thigh + leg)]. Questionnaires (thermal sensation scale: -3 = cold; +3 = hot) will be used to assess participants' thermal comfort/sensation and pain.

ELIGIBILITY:
Inclusion Criteria:

* People with spinal cord injury below thoracic spine 6, at least six months after the injury.
* Healthy adult participants, non-smokers, no disease and/or taking medicines

Exclusion Criteria:

* People under the age of 18;
* People taking any medicines that affect vasomotion (e.g. for hypertension, thrombosis, etc.)
* People with other chronic diseases (e.g. diabetes)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 16 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2020-07-25 (Actual); Study Completion 2020-07-25 (Actual)

PRIMARY OUTCOMES:
Heart rate | 1 hour and 5 minutes
  Heart rate will be continuously monitored using a Polar Team system (Polar® Team 2, Polar Electro Oy, Kempele, Finland
Heart rate variability | 1 hour and 5 minutes
  Heart rate variability will be continuously monitored using a Polar Team system (Polar® Team 2, Polar Electro Oy, Kempele, Finland
Skin temperature | 1 hour and 5 minutes
  Skin temperature (chest, arm, thigh, and leg) will be continuously monitored using iButton sensors type DS1921 H, Maxim/Dallas Semiconductor Corp., USA.
Finger temperature | 1 hour and 5 minutes
  Finger temperature will be monitored throughout baseline and water immersion at 8-s intervals using a data logger (Smartreader 8 Plus, ACR, Vancouver, Canada) interfacing with a computer to allow for their continuous monitoring by the investigators.
Body core temperature | 1 hour and 5 minutes
  Core body temperature will be assessed using telemetric capsules (e-Celsius, BodyCap, Caen, France) that we will give to the participants to ingest prior to the measurement.
Skin blood flow | 1 hour and 5 minutes
  Skin blood flow will be monitored via laser Doppler flowmeter (PeriFlux System 5010, function unit; Perimed, Stockholm, Sweden and PeriFlux System 4002, master unit, satellite unit; Perimed, Stockholm, Sweden)
Change of blood pressure | Change from baseline blood pressure at 10th, 20th, 30th, 40th, 50th and 65th minute.
  Blood pressure will be monitored every 10 minutes with an automatic sphygmomanometer (Omron Healthcare M6 comfort, Japan)
Sweat rate | 1 hour and 5 minutes
  Sweat rate will be measured using a 5.0-cm2 ventilated capsule placed over the forehead and the gastrocnemius. Anhydrous compressed air will be passing through the capsule and over the skin surface (Brooks 5850, mass flow controller, Emerson Electric, Hetfield, PA, USA). The vapor density of the effluent air will be calculating from the relative humidity and temperature measured using the Omega HX93 humidity and temperature sensor (Omega Engineering, Stanford, CT, USA). Sweat rate will be defined as the product of the difference in water content between effluent and influent air and the flow rate. The flow rate through the capsule is 1.13 L min-1. The sweat rate value will be adjusted for skin surface area under the capsule (expressed in mg min-1 cm-2).
Change of thermal comfort | Change from baseline thermal comfort at 10th, 20th, 30th, 40th, 50th and 65th minute.
  Thermal comfort was assessed via the thermal comfort scale (1 = comfortable; 5 = extremely uncomfortable)
Change of thermal sensation | Change from baseline thermal sensation at 10th, 20th, 30th, 40th, 50th and 65th minute.
  Thermal sensation was assessed via the thermal sensation scale (-3 = cold; +3 = hot)

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Flouris, PhD, Study Chair — FAME Laboratory, Department of Exercise Science, University of Thessaly, Greece
Locations (1):
- FAME Lab, Department of Exercise Science, University of Thessaly, Trikala, Thessaly, Greece

IPD SHARING:
Plan to Share IPD: No